CLINICAL TRIAL: NCT04102501
Title: A Randomized, Double-Blind, Controlled, Phase 2/3 Study to Assess Efficacy, Long Term Safety and Tolerability of RT001 in Subjects With Friedreich's Ataxia
Brief Title: A Study to Assess Efficacy, Long Term Safety and Tolerability of RT001 in Subjects With Friedreich's Ataxia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT001-006
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-04

CONDITIONS: Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — RT001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RT001 (Experimental): * 9 capsules daily (8.64 g total dose) given as 3 capsules three times a day (TID) with meals for the first month of treatment.
  * Six capsules daily (5.76 g total dose) given as 3 capsules (BID) with breakfast, and 3 capsules with dinner after the first month of treatment
  Interventions: Drug: RT001
- Placebo (Placebo Comparator): * 9 capsules daily (8.64 g total dose) given as 3 capsules three times a day (TID) with meals for the first month of treatment.
  * Six capsules daily (5.76 g total dose) given as 3 capsules (BID) with breakfast, and 3 capsules with dinner after the first month of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RT001 — RT001 is encapsulated 9-cis, 12-cis-11,11-D2-linoleic acid ethyl ester, which is a site specific (C11) di-deutero synthetic homologue of LA ethyl ester. Each capsule contains 960 mg of RT001.
  Arms: RT001
Drug: Placebo — The placebo product is composed of encapsulated USP safflower oil. The placebo capsules are identical in appearance and size to RT001.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the Efficacy, Long Term Safety and Tolerability of RT001 in subjects with Friedreich's Ataxia

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, tolerability, in subjects with FRDA following the oral administration of study drug (active or placebo capsules). Sixty eligible patients will undergo various assessments at different time points during the the study. The study duration is 13 months which includes screening, treatment and safety follow up phone call.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female 12 to 50 years of age
2. Medical history consistent with the symptoms of FRDA at ≤ 25 years of age
3. Detection of biallelic pathogenic variants in frataxin gene (FXN)
4. Ambulatory (with or without assistive device) and capable of performing other assessments/evaluations.
5. Must be able to walk 25 feet during the timed 1-minute walk

Key Exclusion Criteria:

1. Received treatment with other experimental therapies within the last 30 days prior to the first dose
2. Previously participated in the RT001 trial
3. Refusal to discontinue fish oils or other oil-based supplements for the duration of the study (Screening till last study procedure completed)
4. History of malignancies (other than basal cell carcinomas)
5. Inability to complete CPET protocol
6. Female who is breastfeeding or has a positive pregnancy test
7. History of uncontrolled diabetes mellitus (Type 1 or 2)

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milner, MD, Study Director — Chief Medical Officer
Locations (6):
- United States (6):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - USF Ataxia Research Center, Tampa, Florida
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- RT001: * 9 capsules daily (8.64 g total dose) given as 3 capsules three times a day (TID) with meals for the first month of treatment.
  * Six capsules daily (5.76 g total dose) given as 3 capsules (BID) with breakfast, and 3 capsules with dinner after the first month of treatment
  RT001: RT001 is encapsulated 9-cis, 12-cis-11,11-D2-linoleic acid ethyl ester, which is a site specific (C11) di-deutero synthetic homologue of LA ethyl ester. Each capsule contains 960 mg of RT001.
- Placebo: * 9 capsules daily (8.64 g total dose) given as 3 capsules three times a day (TID) with meals for the first month of treatment.
  * Six capsules daily (5.76 g total dose) given as 3 capsules (BID) with breakfast, and 3 capsules with dinner after the first month of treatment
  Placebo: The placebo product is composed of encapsulated USP safflower oil. The placebo capsules are identical in appearance and size to RT001.
Period: Overall Study
Arm/Group | RT001 | Placebo
Started | 33 | 32
11 Month Visit | 25 | 20
Completed | 25 | 20
Not Completed | 8 | 12
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RT001 | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 13 | 30
  Between 18 and 65 years | 16 | 19 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.0 (5.02) | 21.4 (9.99) | 19.7 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 33
  Male | 19 | 13 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 29 | 59
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 11 Months in Maximum Consumption of Oxygen (mlO2/kg/Min) Using Cardiopulmonary Exercise Testing (CPET)
Description: To measure the change in MVO2 from baseline to Month 11 using CPET
Time Frame: 11 months
Measure: Mean (Standard Error); unit: ml O2/min/kg
Groups:
- RT001; Placebo: Change from Baseline in MVO2 at 11 months
Arm/Group | RT001 | Placebo
Number analyzed (Participants) | 25 | 20
ml O2/min/kg | 0.05 (0.04) | 0.08 (0.04)
Statistical Analysis 1: Comparison: RT001 vs Placebo; Test type: Superiority; p = 0.5858, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in the Timed 1 Minute Walk Distance
Description: Change from baseline Distance walked in 1 minute at 11 months
Time Frame: 11 months
Measure: Mean (Standard Error); unit: inches
Groups:
- RT001: Change from baseline in Timed 1 minute Walk distance
- Placebo: Change from baseline in the timed 1 minute walk distance
Arm/Group | RT001 | Placebo
Number analyzed (Participants) | 25 | 20
inches | -193.83 (73.16) | -220.42 (78.27)
Statistical Analysis 1: Comparison: RT001 vs Placebo; Test type: Superiority; p = 0.8061, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse event reporting was conducted in the ITT population.
Arm/Group | RT001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/32
Other Adverse Events (participants affected / at risk) | 18/33 | 19/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RT001 (N=33) | Placebo (N=32)
non-cardiac chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) — Subject had loss of consciousness due to diabetic ketoacidosis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RT001 (N=33) | Placebo (N=32)
nausea (Gastrointestinal disorders) | 4 (4) | 7 (7)
diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Falls (Injury, poisoning and procedural complications) | 7 (7) | 5 (5)
headache (Nervous system disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT04102501/Prot_SAP_000.pdf